CLINICAL TRIAL: NCT05248386
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Trial to Evaluate the Efficacy and Safety of Intra-articular Injections of RTX-GRT7039 in Adult Subjects With Pain Associated With Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of RTX-GRT7039 in Adult Subjects With Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KF7039-01; 2021-005029-26 (EudraCT Number); U1111-1268-7314 (Other: Universal Trial Number)
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis
Keywords: Knee,; osteoarthritis; pain assessment
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- RTX-GRT7039 (Experimental): Participants will receive intra-articular injections of RTX-GRT7039 during the 52-week double-blind treatment period.
  Interventions: Drug: RTX-GRT7039
- Placebo (Placebo Comparator): Participants will receive intra-articular injections of placebo matching to RTX-GRT7039 during the 52-week double-blind treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RTX-GRT7039 — RTX-GRT7039 intra-articular injection.
  Arms: RTX-GRT7039
Drug: Placebo — Placebo matching RTX-GRT7039 intra-articular injection.
  Arms: Placebo

SUMMARY:
A double-blind, randomized, placebo-controlled, parallel-group, multi-site, clinical trial to confirm the efficacy and safety of repeated injections of RTX-GRT7039 versus placebo in patients who have pain associated with osteoarthritis of the knee despite standard of care.

DETAILED DESCRIPTION:
This trial comprises a total observation period of up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participant has given written informed consent to participate.
* The participant is 18 years of age or older at the Screening Visit.
* The participant has a diagnosis of osteoarthritis of the knee based on American College of Rheumatology criteria and functional capacity class of I to III.
* There is a documented history indicating that participant has insufficient pain relief with previous Standard of Care.

Exclusion Criteria:

* The participant has past joint replacement surgery of the index knee.
* The participant has a history of significant trauma or surgery (e.g., open or arthroscopic) to the index knee within 12 months of Screening.
* The participant has periarticular pain from any cause other than osteoarthritis, including referred pain, bursitis, or tendonitis.
* The participant has clinical hip osteoarthritis on the side of the index knee.
* The participant has pre-existing osteonecrosis, subchondral insufficiency fracture, atrophic osteoarthritis, severe bone on bone osteoarthritis, knee pain attributable to disease other than osteoarthritis, or the participant has rapidly progressing osteoarthritis (RPOA) Type I or Type II.
* The participant has significant malalignment of anatomical axis (medial angle formed by the femur and tibia) of the target knee (varus >10, valgus >10) by X-ray as assessed by independent Central Readers at Screening Visit.
* The participant has other conditions that could affect trial endpoint assessments of the index knee.
* The participant has current clinically significant disease(s) or condition(s) that may affect efficacy or safety assessments, or any other reason which, in the investigator's opinion, may preclude the participant's participation for the full duration of the trial.
* The participant has a history of hypersensitivity to resiniferatoxin (RTX) or any similar component (capsaicin, chili peppers).
* The participant is currently participating or was participating in another investigational drug trial within 3 months prior to the Screening Visit.
* The participant is an employee of the investigator or trial site, with direct involvement in the proposed trial or other trials under the direction of that investigator or trial site or is a family member of the employees or the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (100):
- Canada (7):
  - Cook Street Medical Clinic, Victoria, British Columbia
  - Dr. M. B. Jones, Victoria, British Columbia
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Malton Medical Research, Mississauga, Ontario
  - GRMO (Groupe de Recherche en Rhumatologie et Maladies Osseuses) Inc., Sainte-Foy, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
  - Diex Recherche Victoriaville Inc., Victoriaville, Quebec
- Czechia (14):
  - Lekarna U Svate Anny, Písek, Czech Republic
  - Revmatologie s.r.o., Brno
  - Interni A Revmatologicka Ambulance, Břeclav
  - Vesalion s.r.o., Ostrava
  - Revmatologicka Ambulance, Ostrava
  - Ortopedicko-traumatologicka ambulance, Písek
  - CCBR Czech Prague, s.r.o, Prague
  - CCR Prague, s.r.o, Prague
  - Revmatologicka ambulance, Prague
  - Thomayerova Nemocnice (TN), Prague
  - Fakultni Thomayerova nemocnice s poliklinikou, Prague
  - EUC Klinika, Prague
  - Db Ortopedie s.r.o, Příbram
  - PV-MEDICAL s.r.o. Revmatologicka ambulance, Zlín
- France (8):
  - Centre Hospitalier Universitaire d'Amiens-Picardie - Site Sud, Amiens
  - CHU Amiens Nord, Amiens
  - Hopital Edouard Herriot, Lyon
  - CHU Nimes Cedex, Nîmes
  - Hopital Saint antoine, Paris
  - Cochin Hospital-Paris Descartes University, Paris
  - Hopitaux de Paris (AP-HP) - Groupe Hospitalier Cochin -Assistance Publique, Paris
  - Hopital Lariboisiere,Hospitalier Universitaire Nord, Paris
- Germany (8):
  - Praxis Dr. med. Stephan Grunert, Eichstätt
  - Medizentrum Essen Borbeck, Essen
  - HRF Hamburger Rheuma Forschungszentrum, Hamburg
  - Ortho-Zentrum Karlsruhe, Karlsruhe
  - Velocity Clinical Research Leipzig GmbH, Leipzig
  - AmBeNet, Practice Dr. Dr. med. Hans-Detlev Stahl, Leipzig
  - Centrum fuer Diagnostik und Gesundheit (CDG), München
  - Praxis-Reinfeld-Mitte, Reinfeld
- Italy (5):
  - AOU-Careggi, Florence
  - Universita degli Studi della Campania Luigi Vanvitelli - Azienda Ospedaliera Universitaria, Naples
  - Dipartimento Di Scienze Ortopediche, Traumatologiche, Riabilitative E Plastico-Ricostruttive, Napoli
  - IRCCS Istituto Clinico Humanitas, Rozzano
  - AOU Citta della Salute e della Scienza di Torino, Torino
- Japan (28):
  - Funabashi Municipal Medical Center, Funabashi-shi, Chiba
  - Kamagaya General Hospital, Kamagaya, Chiba
  - Hamanomachi Hospital, Fukuoka, Fukuoka
  - Souseikai Fukuoka Mirai Hospital, Fukuoka, Fukuoka
  - Seiwa-kai medical corporation Hiroshima clinic, Hiroshima, Hiroshima
  - Kosei General Hospital, Mihara, Hiroshima
  - Kosei General Hospital, Mihara-shi, Hiroshima
  - Hakodate Central General Hospital, Hakodate, Hokkaido
  - Sapporo Maruyama Orthopedic Hospital, Sapporo, Hokkaido
  - KKR Sapporo Medical Center, Sapporo, Hokkaido
  - Sapporo kotoni Orthopedies, Sapporo, Hokkaido
  - Kinashi Obayashi Hospital, Takamatsu, Kagawa-ken
  - Japan Organization of Occupational Health and Safety Yokohama Rosai Hospital, Yokohama, Kanagawa
  - Yokohoma Rosai Hospital, Yokohama, Kanagawa
  - Social Medical Care Corporation Hosei-kai Marunouchi Hospital, Nagano, Matsumoto-shi Nagano
  - KKR Tohoku Kosai Hospital, Sendai, Miyagi
  - Nakajo Orthopedic Clinic, Sendai, Miyagi
  - Marunouchi Hospital, Matsumoto, Nagano
  - KKR Tohoku Kosai Hospital, Aoba-ku, Sendai-shi
  - Otsu City Hospital, Ōtsu, Shiga
  - Shimane University Hospital, Izumo, Shimane
  - Japanese Red Cross Hamamatsu Hospital, Hamamatsu, Shizuoka
  - Juntendo University Hospital, Bunkyo-Ku, Tokyo
  - Juntendo University Graduate School of Medicine, Bunkyo-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - Shirahama Hamayu Hospital, Nishimura, Wakayama
  - Juntendo University Hospital, Tokyo
  - Medical Corporation Teda Ooimachi Orthopaedic Surgery and Surgery Clinic, Tokyo
- Mexico (8):
  - Morales Vargas Centro de Investigacion SC, León, Guanajuato
  - Centro Integral en Reumatologia, SA de CV, Guadalajara, Jalisco
  - Clinstile, S.A. de C.V, Cuauhtémoc, Mexico City
  - Consultorio de Reumatologia, Gustavo Adolfo Madero, Mexico City
  - CINTRE, Centro de Investigacion y Tratamiento Reumatologico S.C., Mexico City, Mexico City
  - Dr. Miguel Cortes Hernandez MD, Office of, Cuernavaca, Morelos
  - Centro de Investigacion de Tratamientos Innovadores de Sinaloa S.C., Culiacán, Sinaloa
  - Investigacion y Biomedicina de Chihuahua, Chihuahua City
- Netherlands (3):
  - Medisch Spectrum Twente (MST) - Enschede Haaksbergerstraat, Enschede, KZ
  - PT&R, Beek, Limburg
  - Spaarne Gasthuis (Kennemer Gasthuis), Hoofddorp
- Poland (19):
  - Synexus Poznan Medical Center, Poznan, Greater Poland Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - Reumed Spolka z o.o. Zespol poradni Specjalistycznych Filia Nr 1 Wallenroda, Lublin, Lublin Voivodeship
  - KO-MED Centra Kliniczne Lublin II, Zamość, Lublin Voivodeship
  - Makmed Nzoz, Nadarzyn, Masovian Voivodeship
  - NZOZ Lecznica MAK-MED S.C., Nadarzyn, Masovian Voivodeship
  - Gabinet Internistyczno-Reumatologiczny Piotr Adrian Klimiuk, Bialystok, Podlaskie Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk, Pomeranian Voivodeship
  - INTER CLINIC Piotr Adrian Klimiuk, Bialystok
  - Synexus Gdynia, Gdynia
  - Mazowieckie Centrum Badan Klinicznych, Grodzisk Mazowiecki
  - Synexus Katowice Medical Center, Katowice
  - Centrum Medyczne Pratia Katowice, Katowice
  - Malopolskie Centrum Kliniczne, Krakow
  - St Centrum Medyczne Plejady, Krakow
  - Synexus Polska Sp. z o.o. Oddzial w Lodzi, Lodz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - Synexus Polska Spolka z ograniczona odpowiedzialnoscia Oddzial we Wroclawiu, Wroclaw
  - Centrum Medyczne Kuba-Med Zamosc, Zamość

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Group Web Site (see URL below for details); according to the European Federation of Pharmaceutical Industries and Associations (EFPIA) Data Sharing Principles.
URL: https://www.grunenthal.com/en/research-and-development/clinical-trials/data-sharing-clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- RTX-GRT7039: Participants received intra-articular injections of RTX-GRT7039 (2 injections: Day 1 and Week 26) during the 52-week double-blind treatment period.
  Reporting groups (Full Analysis Set [FAS] and Safety Analysis Set [SAS]) corresponds to all subjects with an Investigational medicinal product (IMP) administration or matching placebo (including incomplete administrations): FAS - based on treatment as randomized (i.e. as planned); SAF - based on treatment received.
- Placebo: Participants received intra-articular injections of placebo matching to RTX-GRT7039 (2 injections: Day 1 and Week 26) during the 52-week double-blind treatment period.
  Reporting groups (Full Analysis Set [FAS] and Safety Analysis Set [SAS]) corresponds to all subjects with an Investigational medicinal product (IMP) administration or matching placebo (including incomplete administrations): FAS - based on treatment as randomized (i.e. as planned); SAF - based on treatment received.
Period: Overall Study
Arm/Group | RTX-GRT7039 | Placebo
Started | 234 | 232
Completed | 202 | 204
Not Completed | 32 | 28
Not completed — Technical problems | 0 | 1
Not completed — Withdrawal by Subject | 15 | 10
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 2 | 4
Not completed — Other | 1 | 0
Not completed — Lack of Efficacy | 14 | 12

BASELINE CHARACTERISTICS:
Population: Reporting groups (Full Analysis Set [FAS] and Safety Analysis Set [SAS]) corresponds to all subjects with an Investigational medicinal product (IMP) administration or matching placebo (including incomplete administrations): FAS - based on treatment as randomized (i.e. as planned); SAF - based on treatment received.
Groups:
- RTX-GRT7039: Participants received intra-articular injections of RTX-GRT7039 (2 injections: Day 1 and Week 26) during the 52-week double-blind treatment period.
- Placebo: Participants received intra-articular injections of placebo matching to RTX-GRT7039 (2 injections: Day 1 and Week 26) during the 52-week double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | RTX-GRT7039 | Placebo | Total
Number analyzed (Participants) | 234 | 232 | 466
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (8.40) | 67.1 (8.32) | 66.8 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 174 | 337
  Male | 71 | 58 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 17 | 33
  Not Hispanic or Latino | 214 | 214 | 428
  Unknown or Not Reported | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean (Standard Error) [LS-mean (SE)] Change From Baseline in WOMAC Pain Subscale Score at Week 12
Description: Difference in mean change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale score at Week 12 in the index knee using an 11-point (0-10) numeric rating scale (NRS) between RTX-GRT7039 and placebo. The WOMAC pain subscale consists of 5 questions using an 11-point numeric rating scale (NRS, from 0 = no pain to 10 = pain as bad as you can imagine).
Time Frame: Baseline up to Week 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | RTX-GRT7039 | Placebo
Number analyzed (Participants) | 234 | 232
score on a scale | -2.959 (0.15) | -2.847 (0.15)

2. Secondary Outcome: LS-mean (SE) Change From Baseline in WOMAC Pain Subscale Score at Week 26
Description: Difference in mean change from baseline in WOMAC pain subscale score at Week 26 in the index knee using an 11-point (0-10) numeric rating scale (NRS) between RTX-GRT7039 and placebo. The WOMAC pain subscale consists of 5 questions using an 11-point numeric rating scale (NRS, from 0 = no pain to 10 = pain as bad as you can imagine).
Time Frame: From Baseline up to Week 26
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | RTX-GRT7039 | Placebo
Number analyzed (Participants) | 234 | 232
score on a scale | -2.564 (0.15) | -2.597 (0.16)

3. Secondary Outcome: LS-mean (SE) Change From Baseline in WOMAC Pain Subscale Score at Week 52
Description: Difference in mean change from baseline in WOMAC pain subscale score at Week 52 in the index knee using an 11-point (0-10) numeric rating scale (NRS) between RTX-GRT7039 and placebo. The WOMAC pain subscale consists of 5 questions using an 11-point numeric rating scale (NRS, from 0 = no pain to 10 = pain as bad as you can imagine).
Time Frame: From Baseline up to Week 52
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | RTX-GRT7039 | Placebo
Number analyzed (Participants) | 234 | 232
score on a scale | -2.686 (0.18) | -2.823 (0.18)

4. Secondary Outcome: LS-mean (SE) Change From Baseline in WOMAC Physical Function Subscale Score at Week 12
Description: Difference in mean change from baseline in WOMAC physical function subscale score at Week 12 in the index knee using an 11-point (0-10) numeric rating scale (NRS) between RTX-GRT7039 and placebo. The WOMAC pain subscale consists of 5 questions using an 11-point numeric rating scale (NRS, from 0 = no pain to 10 = pain as bad as you can imagine).
Time Frame: From Baseline up to Week 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | RTX-GRT7039 | Placebo
Number analyzed (Participants) | 234 | 232
score on a scale | -2.802 (0.14) | -2.740 (0.14)

5. Secondary Outcome: LS-mean (SE) Change From Baseline in WOMAC Physical Function Subscale Score at Week 26
Description: Difference in mean change from baseline in WOMAC physical function subscale score at Week 26 in the index knee using an 11-point (0-10) numeric rating scale (NRS) between RTX-GRT7039 and placebo. The WOMAC pain subscale consists of 5 questions using an 11-point numeric rating scale (NRS, from 0 = no pain to 10 = pain as bad as you can imagine).
Time Frame: From Baseline up to Week 26
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | RTX-GRT7039 | Placebo
Number analyzed (Participants) | 234 | 232
score on a scale | -2.503 (0.14) | -2.552 (0.15)

6. Secondary Outcome: LS-mean (SE) Change From Baseline in WOMAC Physical Function Subscale Score at Week 52
Description: as for outcome 5
Time Frame: From Baseline up to Week 52
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | RTX-GRT7039 | Placebo
Number analyzed (Participants) | 234 | 232
score on a scale | -2.664 (0.16) | -2.728 (0.16)

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Arm/Group | RTX-GRT7039 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/234 | 0/232
Serious Adverse Events (participants affected / at risk) | 17/234 | 14/232
Other Adverse Events (participants affected / at risk) | 53/234 | 40/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RTX-GRT7039 (N=234) | Placebo (N=232)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RTX-GRT7039 (N=234) | Placebo (N=232)
Procedural pain (Injury, poisoning and procedural complications) | 31 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 20
Nasopharyngitis (Infections and infestations) | 10 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results (or parts thereof) of this trial may be published as a publication (e.g., journal publication) or at a congress (e.g., as a poster or presentation). The sponsor reserves the right to review any proposed full publication, poster, or presentation of the results of this trial by the coordinating investigator before they are submitted for publication or public disclosure.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT05248386/Prot_SAP_000.pdf